CLINICAL TRIAL: NCT03642249
Title: Evaluating the Effects of Implementing an Scenario-based Education Initiative and OSCE for Recognition and Management of Delirium in Adult Intensive Care Unit: Randomised Controlled Trial
Brief Title: Education for Recognition and Management of Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N201803104
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2019-09

CONDITIONS: Delirium; Intensive Care Unit Syndrome; Nurse-Patient Relations
Keywords: delirium; knowledge translation; Objective Structured Clinical Examination; evidence-based practice
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration); and
  3. delirium care OSCE and reflective activity (30 minutes in duration).
  Interventions: Behavioral: OSCEs; Behavioral: Lecture; Behavioral: E-learning
- control group (Active Comparator): 1. face-to-face delirium care session (30 minutes in duration);
  2. online learning delirium care activities (20 minutes in duration)
  Interventions: Behavioral: Lecture; Behavioral: E-learning

INTERVENTIONS:
Behavioral: OSCEs — Scenario-based education intervention, including objective structured clinical examinations (OSCEs)
  Arms: experimental group
Behavioral: Lecture — Face-to-face Education using Delirium Care Flip Chart
Behavioral: E-learning — delirium care video

SUMMARY:
Delirium is a disturbance in consciousness with reduced ability to focus, sustain, or shift attention that occurs over a short period of time and tends to fluctuate over the course of the day. 50% to 81.7% had delirium during their ICU hospitalization. Delirium is associated with increased physical restraint, ventilation use, length of ICU stay, and mortality. However, there is no established delirium care pathway in target hospital. Chen et al. (2014) demonstrated that structured assessment stations with immediate feedback may improve overall learning efficiency over an EBP workshop alone. However, no published delirium care education study has used OSCEs as an intervention for healthcare professionals. The aim is to evaluate the effects of implementing a Scenario-based education intervention, including objective structured clinical examinations (OSCEs) on delirium care among healthcare professionals. This is a knowledge translation research, builds on eight years of delirium care research in University of Wollongong, Australia. The research will be undertaken at ICUs in a medical center in northern of Taiwan. There are two phases: (1) systematic review to identify delirium screen tool, and (2) a randomized controlled trial was conducted to determine the effects of implementing a Scenario-based education intervention, including OSCE (experimental group), and on-line education only (control group) focused on recognition and management of delirium. The hypothesis is: Scenario-based education intervention, including OSCE can increase the competence and self-efficacy among healthcare professionals in delirium care.

DETAILED DESCRIPTION:
OSCEs are an integral aspect of all levels of medical education but limited to undergraduate nursing and allied health education. OSCEs are rarely used in the workplace as learning activities with nursing and allied health clinicians. This is the reason why this education initiative was innovative. OSCEs are simulated 'real life' clinical scenarios presented to clinicians who are required to demonstrate to an assessor the clinical tasks which form an OSCE scenario.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurse worked in acute care unit and care with critical patients
* Age > 20 years old.

Exclusion Criteria:

* Unwilling to involved the research

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Delirium Knowledge and Skills at the time Immediately after the intervention and Six weeks | T0(Baseline), T1(Immediately after the intervention), T2(Six weeks after the intervention)
  Delirium Knowledge and Skills Test (included 18 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Kee-Hsin Chen, PhD, Study Director — Taipei Medical University
Locations (1):
- Wan Fang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellelli G, Morandi A, Davis DH, Mazzola P, Turco R, Gentile S, Ryan T, Cash H, Guerini F, Torpilliesi T, Del Santo F, Trabucchi M, Annoni G, Maclullich AM. Corrigendum to 'Validation of the 4AT, a new instrument for rapid delirium screening: a study in 234 hospitalised older people'. Age Ageing. 2015 Jan;44(1):175. doi: 10.1093/ageing/afu181. No abstract available. PMID 25477307
- [Background] Campbell N, Boustani MA, Ayub A, Fox GC, Munger SL, Ott C, Guzman O, Farber M, Ademuyiwa A, Singh R. Pharmacological management of delirium in hospitalized adults--a systematic evidence review. J Gen Intern Med. 2009 Jul;24(7):848-53. doi: 10.1007/s11606-009-0996-7. Epub 2009 May 8. PMID 19424763
- [Background] Coyle H, Traynor V, Solowij N. Computerized and virtual reality cognitive training for individuals at high risk of cognitive decline: systematic review of the literature. Am J Geriatr Psychiatry. 2015 Apr;23(4):335-359. doi: 10.1016/j.jagp.2014.04.009. Epub 2014 May 14. PMID 24998488
- [Background] Coyle MA, Burns P, Traynor V. Is it My Job? The Role of RNs in the Assessment and Identification of Delirium in Hospitalized Older Adults: An Exploratory Qualitative Study. J Gerontol Nurs. 2017 Apr 1;43(4):29-37. doi: 10.3928/00989134-20170111-02. Epub 2017 Jan 18. PMID 28095583
- [Background] De J, Wand APF, Smerdely PI, Hunt GE. Validating the 4A's test in screening for delirium in a culturally diverse geriatric inpatient population. Int J Geriatr Psychiatry. 2017 Dec;32(12):1322-1329. doi: 10.1002/gps.4615. Epub 2016 Oct 20. PMID 27766672
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fox MT, Persaud M, Maimets I, Brooks D, O'Brien K, Tregunno D. Effectiveness of early discharge planning in acutely ill or injured hospitalized older adults: a systematic review and meta-analysis. BMC Geriatr. 2013 Jul 6;13:70. doi: 10.1186/1471-2318-13-70. PMID 23829698
- [Background] Han JH, Wilson A, Graves AJ, Shintani A, Schnelle JF, Dittus RS, Powers JS, Vernon J, Storrow AB, Ely EW. Validation of the Confusion Assessment Method for the Intensive Care Unit in older emergency department patients. Acad Emerg Med. 2014 Feb;21(2):180-7. doi: 10.1111/acem.12309. PMID 24673674
- [Background] Hsu LL, Huang YH, Hsieh SI. The effects of scenario-based communication training on nurses' communication competence and self-efficacy and myocardial infarction knowledge. Patient Educ Couns. 2014 Jun;95(3):356-64. doi: 10.1016/j.pec.2014.03.010. Epub 2014 Mar 20. PMID 24718019
- [Background] Hu RF, Jiang XY, Chen J, Zeng Z, Chen XY, Li Y, Huining X, Evans DJ. Non-pharmacological interventions for sleep promotion in the intensive care unit. Cochrane Database Syst Rev. 2015 Oct 6;2015(10):CD008808. doi: 10.1002/14651858.CD008808.pub2. PMID 26439374
- [Background] Inouye SK, Bogardus ST Jr, Charpentier PA, Leo-Summers L, Acampora D, Holford TR, Cooney LM Jr. A multicomponent intervention to prevent delirium in hospitalized older patients. N Engl J Med. 1999 Mar 4;340(9):669-76. doi: 10.1056/NEJM199903043400901. PMID 10053175
- [Background] Kuladee S, Prachason T. Development and validation of the Thai version of the 4 'A's Test for delirium screening in hospitalized elderly patients with acute medical illnesses. Neuropsychiatr Dis Treat. 2016 Feb 24;12:437-43. doi: 10.2147/NDT.S97228. eCollection 2016. PMID 26966365
- [Background] Lahariya S, Grover S, Bagga S, Sharma A. Delirium in patients admitted to a cardiac intensive care unit with cardiac emergencies in a developing country: incidence, prevalence, risk factor and outcome. Gen Hosp Psychiatry. 2014 Mar-Apr;36(2):156-64. doi: 10.1016/j.genhosppsych.2013.10.010. Epub 2013 Oct 16. PMID 24295565
- [Background] O'Sullivan D, Brady N, Manning E, O'Shea E, O'Grady S, O 'Regan N, Timmons S. Validation of the 6-Item Cognitive Impairment Test and the 4AT test for combined delirium and dementia screening in older Emergency Department attendees. Age Ageing. 2018 Jan 1;47(1):61-68. doi: 10.1093/ageing/afx149. PMID 28985260
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Pierre RB, Wierenga A, Barton M, Branday JM, Christie CD. Student evaluation of an OSCE in paediatrics at the University of the West Indies, Jamaica. BMC Med Educ. 2004 Oct 16;4:22. doi: 10.1186/1472-6920-4-22. PMID 15488152
- [Background] Salluh JI, Wang H, Schneider EB, Nagaraja N, Yenokyan G, Damluji A, Serafim RB, Stevens RD. Outcome of delirium in critically ill patients: systematic review and meta-analysis. BMJ. 2015 Jun 3;350:h2538. doi: 10.1136/bmj.h2538. PMID 26041151
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Tamune H, Yasugi D. How can we identify patients with delirium in the emergency department?: A review of available screening and diagnostic tools. Am J Emerg Med. 2017 Sep;35(9):1332-1334. doi: 10.1016/j.ajem.2017.05.026. Epub 2017 May 22. PMID 28571901
- [Background] Traynor V, Inoue K, Crookes P. Literature review: understanding nursing competence in dementia care. J Clin Nurs. 2011 Jul;20(13-14):1948-60. doi: 10.1111/j.1365-2702.2010.03511.x. Epub 2011 Mar 15. PMID 21401762
- [Background] Wong CL, Holroyd-Leduc J, Simel DL, Straus SE. Does this patient have delirium?: value of bedside instruments. JAMA. 2010 Aug 18;304(7):779-86. doi: 10.1001/jama.2010.1182. PMID 20716741
- [Background] Ytterberg SR, Harris IB, Allen SS, Anderson DC, Kofron PM, Kvasnicka JH, McCord JP, Moller JH. Clinical confidence and skills of medical students: use of an OSCE to enhance confidence in clinical skills. Acad Med. 1998 Oct;73(10 Suppl):S103-5. doi: 10.1097/00001888-199810000-00060. No abstract available. PMID 9795667
- [Background] Zaal IJ, Slooter AJ. Delirium in critically ill patients: epidemiology, pathophysiology, diagnosis and management. Drugs. 2012 Jul 30;72(11):1457-71. doi: 10.2165/11635520-000000000-00000. PMID 22804788